CLINICAL TRIAL: NCT02626689
Title: Burden of Beta-Thalassemia - Quality of Life and Health Care Resource Utilization- A Prospective Observational Study
Brief Title: To Document the Burden of Illness on the Quality of Life and the Impact on Healthcare Utilization in (Beta) β-thalassemia Subjects Who Are Transfusion Dependent (TD) and Non-transfusion Dependent (NTD) Receiving Standard of Care
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: ACE-536-B-THAL-003
Record Dates: First submitted 2015-11-05; First posted 2015-12-10 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-04

CONDITIONS: Beta-Thalassemia
Keywords: Beta-Thalassemia; Quality of Life; Healthcare Utilization; Transfusion dependent (TD) β-thalassemia; Non-transfusion dependent β-thalassemia; Standard of care; TransQoL; SF36v2; Fact-An; NTD beta-thalassemia PRO
MeSH Terms: conditions — beta-Thalassemia | interventions — Quality of Life; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- β-thalassemia transfusion dependent subjects: Participants will complete 3 quality of life instruments (i.e. FACT-AN, the SF-36v2, and the TranQol) once every 3 weeks, in addition to a TranQol instrument on the day of a RBC transfusion. Continuous monitoring of Healthcare Resource Utilization will be conducted throughout the course of the study at each clinical visit.
  Interventions: Other: Quality of Life (QOL) questionnaires; Other: Healthcare Resource Utilization
- β-thalassemia Non Transfusion Dependent (NTD) subjects: Participants will complete 2 quality of life instruments (i.e. FACT-An and the the SF-36v2l) once every 3 weeks, in addition to completing the non-transfusion dependent Patient Recorded Outcome (PRO) tool on a daily basis. Continuous monitoring of Healthcare Resource Utilization will be conducted throughout the course of the study at each clinical visit.
  Interventions: Other: Quality of Life (QOL) questionnaires; Other: Healthcare Resource Utilization

INTERVENTIONS:
Other: Quality of Life (QOL) questionnaires — Monitoring of FACT-AN, SF-36V2, TransQol, and NTD PRO assessments,
Other: Healthcare Resource Utilization — Monitoring and reviewing HealthCare Resource Utilization information.

SUMMARY:
This is a multi-site, prospective, observational study implemented in β-thalassemia treatment centers from 5 countries (Italy, Turkey, Greece, Lebanon, and Thailand). Approximately one to two study sites will be identified per country and approximately 20 β-thalassemia subjects will be enrolled per country (10 transfusion dependent (TD) and 10 Non-transfusion dependent (NTD) with a total of approximately 100 subjects. This study will not interfere with or influence the routine clinical management of β-thalassemia patients. Outcomes of interest will be collected prospectively for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

For the transfusion dependent (TD) subjects:

1. Male or female, >18 years of age at the time of signing the informed consent document (ICF);
2. Documented diagnosis of β-thalassemia or hemoglobin E/ β-thalassemia;
3. TD - defined as: ≥6 Red Blood Cells (RBC) units in the 24 weeks prior to study participation and no transfusion free period for ≥35 days during that period; and
4. Performance status: Eastern Cooperative Oncology Group (ECOG) score of 0 to 1.

For the non-transfusion dependent (NTD) subpopulation

1. Male or female, >18 years of age at the time of signing the informed consent document (ICF).
2. Documented diagnosis of β-thalassemia or hemoglobin E/ β-thalassemia
3. NTD - defined as: 0 to 5 RBC units received during the 24-week period prior to study participation (not including RBC transfusions units administered for elective surgery);
4. Most recent hemoglobin ≤10 g/dL (hemoglobin values ≤ 21 days post-transfusion will be excluded)
5. Performance status: ECOG score of 0 to 1.

Exclusion Criteria:

For TD Subpopulation:

1. A diagnosis of hemoglobin S/β-thalassemia;
2. Any significant psychiatric or medical conditions not related to thalassemia that would prevent the subject from participating in the study;
3. Inability to read or understand the local official languages; or
4. Participated in another clinical trial (interventional) <30 days prior to study participation

For NTD Subpopulation:

1. Received RBC transfusion ≤ 8 weeks prior to study enrollment;
2. A diagnosis of hemoglobin S/β-thalassemia;
3. Any significant psychiatric or medical conditions not related to thalassemia that would prevent the subject from participating in the study;
4. Inability to read or understand the local official languages; or
5. Participated in another clinical trial (interventional) <30 days prior to study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: β-thalassemia subjects who are transfusion dependent (TD) and non-transfusion dependent (NTD)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-01-03 (Actual); Study Completion 2017-01-03 (Actual)

PRIMARY OUTCOMES:
Change in the Physical component score (PSC) over the study period versus the country specific population norms using the 36-item Short Form (SF-36) Quality of Life instrument | Up to 6 months
  Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.
Change in the Mental component score (MCS) over the study period versus the country specific population norms using the 36-item Short Form (SF-36) Quality of Life instrument | Up to 6 months
  Short Form 36-Item Health Survey, Version 2 (SF-36) is a self-administered instrument that measures the impact of disease on overall quality of life and consists of 36 questions in eight domains (physical function, pain, general and mental health, vitality, social function, physical and emotional health). Norm-based scores were used in analyses, calibrated so that 50 is the average score and the standard deviation equals 10. Higher scores indicate a higher level of functioning. The physical functioning domain assesses limitations in physical activities because of health problems. A positive change from Baseline score indicates an improvement.

SECONDARY OUTCOMES:
Change in the total scores over the study period using the The Functional Assessment of Cancer Therapy-Anemia (FACT-An) questionnaire | Up to 6 months
  The FACT-An questionaire is used to assess leath-related quality of life (HRQol). It measures the impact of fatigue and other anemia-related symptoms on patient functioning. The overall score range for the FACT-An is 0-188. Higher scores indicate better HRQoL. In addition to general HRQoL, the FACT-An measures the impact of fatigue and other anemia-related symptoms on patient functioning. Patients with higher hemoglobin levels and better performance status reported significantly higher scores on these instruments (including the newly created subscales) than did those with lower hemoglobin levels and poorer performance status
Change in the total scores over the study period using the Tran-QOL questionnaire | Up to 6 months
  The Tran Qol is a new disease specific QOL measure for adults with B-Thalassemia with a score ranging from 0-100. It measures the quality of life issues of patients with B-Thalassemia by assessing physical health, emotional health, family functioning and school/career functioning. Higher scores indicate better health related quality of life (HRQOL). A positive change from baseline indicates an improvement in overall HRQol.
Change in the total scores over the study period using the Patient Reported Outcome (PRO) questionnaire in non-transfusion dependent (NTD) subjects | Up to 6 months
  For NTD subjects, they will complete a Patient Reported Outcome (PRO) PRO via e-diary each evening before bedtime. For all subjects, physical activities will be recorded continuously via Fitbit for the entire study period.
Changes in the annual Healthcare Resource Care (HRC) involving the number of office visits | Up to 6 months
  Healthcare resource utilization will be measured by the number of office visits a B-thal patient has over the course of 6 months while involved in the study.
Number of minutes spent in sedentary, lightly active, fairly active, or very active lifestyles | Up to 6 months
  Number of minutes a patient will spend in sedentary, lightly active, fairly active, and very active levels.
Changes in the annual Healthcare Resource Care (HRC) involving the number of prescriptions dispensed | Up to 6 months
  Healthcare resource utilization will be measured by the number of prescriptions dispensed for a B-thal patient over the course of 6 months while involved in the study
Changes in the annual Healthcare Resource Care (HRC) involving the number of procedures undergone | Up to 6 months
  Healthcare resource utilization will be measured by the number of procedures undergone for a B-thal patient over the course of 6 months while involved in the study
Changes in the annual Healthcare Resource Care (HRC) involving the number of lab assessments completed | Up to 6 months
  Healthcare resource utilization will be measured by the number of lab assessments completed for a B-thal patient over the course of 6 months while involved in the study, relating to the following lab assessments: hematology, clinical chemistry, renal, hepatic, iron parameters, endocrine parameters, and urinalysis.
Changes in the annual Healthcare Resource Care (HRC) involving the number of days that a patient is hospitalized | Up to 6 months
  Healthcare resource utilization will be measured by the number of days the B-thal patient was hospitalized over the course of 6 months while involved with the study, including the number of days that the patient was in the Intensive Care Unit (ICU)
Changes in the annual Healthcare Resource Care (HRC) involving the number of emergency room visits | Up to 6 months
  Healthcare resource utilization will be measured by the number of emergency room visits the B-thal patient had over the course of the 6 months while involved with the study
Percentage of time spent in sedentary, lightly active, fairly active, or very active lifestyles | Up to 6 months
  Percentage of time a patient will spend in sedentary, lightly active, fairly active, or very active lifestyles

CONTACTS AND LOCATIONS:
Overall Officials: Xiaohan (Henry) HU, MD, MPH, PhD, Study Director — Celgene
Locations (5):
- Aghia Sofia Children's Hosptial, Athens, Goudi, Greece
- Fondazione IRCCS Ca Granda Ospedale Maggiore, Milan, Italy
- American University of Beirut Medical Center, Beirut, Lebanon
- Faculty of Medicine Siriraj Hospital, Mahidol University, Bangkok, Bangkoknoi, Thailand
- Cukurova University Medical Faculty Balcali Hospital, Çukurova, Turkey (Türkiye)